CLINICAL TRIAL: NCT07082920
Title: A Phase 1b Study of JNJ-78278343, a T-cell Redirecting Agent Targeting Human Kallikrein 2 (KLK2), in Combination With JNJ-95298177, an Antibody Drug Conjugate Targeting Prostate Specific Membrane Antigen, for Prostate Cancer
Brief Title: A Study of JNJ-78278343 in Combination With JNJ-95298177 for Treatment of Prostate Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 78278343PBPCR1004
Record Dates: First submitted 2025-07-22; First posted 2025-07-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Confirmation (Experimental): Participants will receive JNJ-78278343 in combination with JNJ-95298177 in a dose de-escalation schedule in accordance with the Bayesian Optimal Interval Design (BOIN) design to determine the recommended phase 2 combination dose (RP2CD) regimen.
  Interventions: Drug: JNJ-78278343; Drug: JNJ-95298177
- Part 2: Dose Expansion (Experimental): Participants will receive JNJ-78278343 in combination with JNJ-95298177 at the RP2CD as determined in Part 1 of the study to confirm the safety and anti-tumor activity.
  Interventions: Drug: JNJ-78278343; Drug: JNJ-95298177

INTERVENTIONS:
Drug: JNJ-78278343 — JNJ-78278343 will be administered intravenously.
  Other Names: Pasritamig
Drug: JNJ-95298177 — JNJ-95298177 will be administered intravenously.
  Other Names: ARX517

SUMMARY:
The purpose of this study is to identify the recommended phase 2 combination dose (RP2CD) of JNJ-78278343 in combination with JNJ-95298177 in Part 1 (Dose confirmation) of the study and to determine how safe and tolerable the RP2CD is for treatment of participants with metastatic castration-resistant prostate cancer (mCRPC; a stage of prostate cancer where the cancer has spread beyond the prostate and is resistant to hormonal therapy) in Part 2 (Dose expansion) of study.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the prostate. Primary small cell carcinoma, carcinoid tumor, neuroendocrine (NE) carcinoma, or large cell NE carcinoma arising in the prostate are not allowed; however, adenocarcinomas with NE features (for example [e.g.], immunohistochemistry [IHC] with both androgen receptor [AR]- and NE-marker positivity) are allowed
* Must have metastatic castration-resistant prostate cancer (mCRPC)
* PSA must measure at least 2 nanograms per milliliters (ng/mL) at screening
* Measurable or evaluable disease
* Prior orchiectomy or medical castration; or, for participants who have not undergone orchiectomy, must be receiving ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analog (agonist or antagonist) prior to the first dose of study drug and must continue this therapy throughout the treatment phase
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1

Exclusion criteria:

* Toxicity related to prior anticancer therapy that has not returned to grade less than or equal to (<=) 1 or baseline levels (except for alopecia and vitiligo)
* Known allergies, hypersensitivity, or intolerance to any of the components (e.g., excipients) of JNJ-78278343 or JNJ-95298177
* Participants with leptomeningeal disease or brain metastases, with the exception of participants with definitively, locally treated brain metastases that are clinically stable and asymptomatic greater than (>) 2 weeks, and who are off corticosteroid treatment for at least 2 weeks prior to first dose of study treatment
* Treatment with any anti-cancer or investigational agents within 14 days prior to the first dose of study treatment; specific requirements for certain anti-cancer therapies are as follows:

  1. Any T-cell redirecting treatment (e.g., CD3-directed bispecific or Chimeric Antigen Receptor T-cell [CAR-T] therapy) within 90 days prior to the first dose of study treatment
  2. Immune checkpoint inhibitors within 6 weeks prior to the first dose of study treatment
  3. Radium (Ra) 223 dichloride within 28 days prior to the first dose of study treatment
  4. Any prior treatment with kallikrein-related peptidase 2 (KLK2)-targeted therapy
  5. Any prior prostate-specific membrane antigen (PSMA)-targeting therapy (that is [i.e.], participants who received PSMA-targeting radioconjugates are excluded) [Parts 2A and 2B only]. Prior PSMA RLT is allowed in Part 1 and required for Part 2C and Part 2D but last dose must be >3 months prior to the first dose of study treatment
  6. Any prior antibody drug conjugates (ADCs) with microtubule inhibitor payloads (e.g., auristatins, maytansinoids, tubulysins)
* Any serious underlying medical conditions or other issue that would impair the ability of the participant to receive or tolerate the planned treatment at the investigational site to understand the informed consent, or any condition for which, in the opinion of the investigator, participation would not be in the best interest of the participant or that could prevent, limit, or confound the protocol-specified assessments

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) by Severity | Up to 2 years 2 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/biological agent under study. Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event. Cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity syndrome (ICANS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines and ocular events will be graded using the alternative scale provided in the protocol.
Part 1: Number of Participants With Dose-Limiting Toxicity (DLT) | Up To Day 22
  High grade hematologic or non-hematologic toxicities with exceptions and/or toxicities leading to treatment discontinuation will be regarded as DLT.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years 2 months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to the response evaluation criteria in solid tumors (RECIST) version 1.1 response criteria without evidence of bone progression according to prostate cancer working group 3 (PCWG3).
Prostate-Specific Antigen (PSA) Response Rate | Up to 2 years 2 months
  PSA response rate is defined as the percentage of participants with a decline of PSA of 50% or more from baseline.
Radiographic Progression-Free Survival (rPFS) | Up to 2 years 2 months
  rPFS is defined as the time from the date of first dose of JNJ-78278343 or JNJ-95298177 until the date of radiographic disease progression or death, whichever comes first.
Time to Response (TTR) | Up to 2 years 2 months
  TTR is defined for the responders as the time from the date of first dose of any study treatment to the date of first documented response.
Duration of Response (DOR) | Up to 2 years 2 months
  DOR will be calculated among responders (PR or better) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3 or RECIST version 1.1 response criteria, or death due to any cause, whichever occurs first.
Serum Concentration of JNJ-78278343 | Up to 2 years 2 months
  Serum samples will be analyzed to determine concentrations of JNJ-78278343.
Serum Concentration of JNJ-95298177 | Up to 2 years 2 months
  Serum samples will be analyzed to determine concentrations of JNJ-95298177 (including ADC, total antibody and payload pAF-AS269).
Number of Participants With Anti-JNJ-78278343 Antibodies | Up to 2 years 2 months
  Serum samples will be analyzed for the detection of anti-JNJ-78278343 antibodies using a validated assay method.
Number of Participants With Anti-JNJ-95298177 Antibodies | Up to 2 years 2 months
  Serum samples will be analyzed for the detection of anti-JNJ-95298177 antibodies using a validated assay method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical trial, Study Director — Janssen Research & Development, LLC
Locations (6):
- United States (4):
  - Florida Cancer Specialists, Sarasota, Florida
  - Columbia University Medical Center, New York, New York
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Fred Hutchinson Cancer Center, Seattle, Washington
- United Kingdom (2):
  - The Christie Nhs Foundation Trust, Manchester
  - Royal Marsden Hospital (Sutton), Sutton

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency